CLINICAL TRIAL: NCT06146101
Title: A Phase II/III, Randomised, Double-Blind Clinical Trial to Determine the Safety and Efficacy of IHL-42X in Subjects With Obstructive Sleep Apnoea Who Are Intolerant, Non-Compliant, or Naïve to Positive Airway Pressure
Brief Title: RePOSA-Revealing the Efficacy of IHL-42X Use in Patients With OSA
Acronym: REPOSA
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Incannex Healthcare Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IHL42XOSAP2/3; U1111-1302-4915 (Other: WHO)
Record Dates: First submitted 2023-11-17; First posted 2023-11-24 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-02

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Dronabinol; Acetazolamide

STUDY DESIGN:
Intervention Model Description: Phase 2 (3 arms)
  1. IHL-42X low dose (2.5mg dronabinol, 125mg acetazolamide)
  2. IHL-42X high dose (5mg dronabinol, 250mg acetazolamide)
  3. Placebo
  Phase 3 (4 Arms)
  1. IHL-42X (Optimal dose from phase 2)
  2. Dronabinol (equivalent dose strength to that in the IHL-42X optimal dose strength)
  3. Acetazolamide (equivalent dose strength to that in the IHL-42X optimal dose strength)
  4. Placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (7):
- Phase 2 Investigational Product - IHL-42X Low dose (Experimental): IHL-42X (2.5 mg dronabinol + 125 mg acetazolamide), one capsule self-administered once daily every night approximately 1 hour prior to bed for 4 weeks.
  Interventions: Drug: IHL-42X Low Dose
- Phase 2 Investigational Product - IHL-42X High dose (Experimental): IHL-42X (5 mg dronabinol + 250 mg acetazolamide), one capsule self-administered once daily every night approximately 1 hour prior to bed for 4 weeks.
  Interventions: Drug: IHL-42X High Dose
- Phase 2 Placebo (Placebo Comparator): One capsule self-administered once daily every night approximately 1 hour prior to bed for 4 weeks.
  Interventions: Drug: Placebo
- Phase 3 Investigational Product - IHL-42X (Experimental): IHL-42X (dose will be identified based on the safety and efficacy results in Phase II), one capsule self-administered once daily every night approximately 1 hour prior to bed for 52 weeks.
  Interventions: Drug: IHL-42X (Optimal Dose)
- Phase 3 Comparator - Reference Listed Drug/Dronabinol (Active Comparator): One capsule of dronabinol (equivalent dose strength to that in the IHL-42X optimal dose strength) self-administered once daily every night approximately 1 hour prior to bed for 3 months then IHL-42X (optimal dose) one capsule self-administered once daily every night approximately 1 hour prior to bed for the remaining 9 months.
  Interventions: Drug: Dronabinol
- Phase 3 Comparator - Reference Listed Drug/Acetazolamide (Active Comparator): One capsule of acetazolamide (equivalent dose strength to that in the IHL-42X optimal dose strength) self-administered once daily every night approximately 1 hour prior to bed for 3 months then IHL-42X (optimal dose) one capsule self-administered once daily every night approximately 1 hour prior to bed for the remaining 9 months.
  Interventions: Drug: Acetazolamide
- Phase 3 Placebo (Placebo Comparator): One capsule self-administered once daily every night approximately 1 hour prior to bed for 52 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IHL-42X Low Dose — Softgel capsule
  Other Names: Phase 2 Investigational Product - IHL-42X Low dose
  Arms: Phase 2 Investigational Product - IHL-42X Low dose
Drug: IHL-42X High Dose — Softgel capsule
  Other Names: Phase 2 Investigational Product - IHL-42X High dose
  Arms: Phase 2 Investigational Product - IHL-42X High dose
Drug: Placebo — Softgel capsule
  Other Names: Phase 2 Placebo
  Arms: Phase 2 Placebo
Drug: IHL-42X (Optimal Dose) — Softgel capsule
  Other Names: Phase 3 Investigational Product - IHL-42X
  Arms: Phase 3 Investigational Product - IHL-42X
Drug: Dronabinol — Softgel capsule
  Other Names: Phase 3 Comparator - Reference Listed Drug/Dronabinol
  Arms: Phase 3 Comparator - Reference Listed Drug/Dronabinol
Drug: Acetazolamide — Softgel capsule
  Other Names: Phase 3 Comparator - Reference Listed Drug/Acetazolamide
  Arms: Phase 3 Comparator - Reference Listed Drug/Acetazolamide
Drug: Placebo — Softgel capsule
  Other Names: Phase 3 Placebo
  Arms: Phase 3 Placebo

SUMMARY:
The goal of this randomised, double-blind phase II/III clinical trial is to determine the safety and efficacy of IHL-42X in subjects with obstructive sleep apnoea who are intolerant, non-compliant, or naïve to positive airway pressure.

Phase II study will be a 4-week dose-finding study comparing two dose strengths of IHL-42X to placebo. The optimal dose strength will be selected based on comparing the safety and efficacy of the two IHL-42X dose strengths to placebo over a 4-week treatment period. The three treatment groups are; IHL-42X Low dose (2.5mg dronabinol, 125mg acetazolamide), IHL-42X High dose (5mg dronabinol, 250mg acetazolamide) and Placebo. Each treatment group will enrol approximately 40 patients per treatment arm, for a total of approximately 120 patients.

The safety and efficacy results of the Phase II study will be used to select the dose strength of IHL-42X and corresponding doses of dronabinol and acetazolamide in Phase III.

Phase III study will use the optimal dose strength of IHL-42X identified in Phase II and will be compared to the component active pharmaceutical ingredients at equivalent dose strengths to those found in the IHL-42X optimal dose strength and placebo over 52 weeks. The four treatment groups are; IHL-42X (optimal dose from Phase II), Acetazolamide (equivalent dose strength to that in the IHL-42X optimal dose strength), Dronabinol (equivalent dose strength to that in the IHL-42X optimal dose strength) and placebo. The treatment groups will enrol approximately 165 patients in IHL-42X, approximately 55 patients in dronabinol, approximately 55 in acetazolamide, and approximately 165 in placebo, for a total of approximately 440 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years of age
2. Screening polysomnography (PSG) findings confirmed on central over-read:

   1. AHI ≥15
   2. ≤ 25% central or mixed apneas/hypopneas
   3. no Cheyne-Stokes respiration
   4. total sleep time ≥ 2 hours
3. Intolerant, non-compliant, or naïve to PAP (Note: No more than 25% of the study population will consist of PAP-naïve patients). Patients will be identified as intolerant, non-compliant, or naïve to PAP devices by the following criteria:

   1. Patients are regarded as PAP-non-compliant if they do not use PAP for ≥ 4 hours for at least 21 nights during consecutive 30-day period based on data collected from the PAP device (eg, SD storage cards) and/or a cloud-based repository of PAP device data.
   2. Patients are regarded as PAP-intolerant if they are former PAP users, ie, a PAP device that they have not used for >30 days or who do not have access to PAP device
   3. Patients are regarded as PAP-naïve if they have no prior experience with PAP. Patients who have undergone a split-study, ie, a study of PAP during PSG, are not considered PAP- naïve and should be categorised according to a through b above. (Note: PAP-naïve patients will have the benefits and risks of PAP explained at screening, including that PAP is standard of care for OSA. These patients also have the option to withdraw from the study at any time if he/she elects to be treated with PAP or other alternative therapy such as an oral appliance or surgery)
4. Must agree not to take any form of cannabis or cannabinoid, or any other illicit or recreational drug with the exception of the investigational product (IP) while participating in this study.
5. A female patient of childbearing potential must agree to use 2 approved methods of contraception. Approved methods of contraception include the following:

   1. Intra-uterine device in place for at least 3 months prior to Day 1 through to 10 days following the last dose of the study drug
   2. Barrier method (condom or diaphragm) for at least 3 months prior to Day 1 through to 10 days after the last dose of the study drug
   3. Stable hormonal contraceptive which includes oral, intravaginal, intrauterine, transdermal, injectable, or implantable methods of hormonal contraception for at least 3 months prior to Day 1.

   A female will not be considered of childbearing potential if:
   1. 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum FSH levels > 40 mIU/ml
   2. undergone bilateral tubal ligation, hysterectomy, or bilateral oophorectomy at least 6 months prior to Day 1
6. A male patient must agree to use at least 1 approved method of contraception (or as required by local regulations) while engaging in sexual activity from study Day -1 through End-of-Study (EOS) follow-up and/or up to 10 days following the last administration of the study drug. Male patients must not donate sperm during this same period. Approved methods of contraception include the following:

   1. Barrier method (condom) for at least 14 days prior to Day 1 through to 10 days after the final dose of the study drug
   2. Surgical sterilisation (vasectomy) at least 6 months prior to Day 1
7. Voluntarily written consent to participate in the study and be willing and able to participate in all scheduled visits, treatment plans, tests, and other study procedures according to the protocol

Exclusion Criteria:

1. Body mass index >45 kg/m2
2. PAP-compliant, defined by the use of PAP for ≥ 4 hours for at least 21 nights during the consecutive 30-day period
3. Current use of oral appliances (eg, mandibular advancement device, tongue retaining device, or mouth guard)
4. Maxillomandibular advancement, upper airway, or bariatric surgery within the last 6 months prior to first administration of the study drug; or patients who are considering surgical treatment
5. Use of benzodiazepines, sedative-hypnotics, or stimulants (ATC N06B, N05C, N05BA, N03AE, and N01AF categories) to treat insomnia, OSA, other sleep disorders
6. Pierre Robin, Treacher Collins, or other craniofacial malformation syndrome, or grade ≥3 tonsillar hypertrophy
7. Chronic neuromuscular disorders such as motor neuron disease, muscular dystrophy, or myopathy
8. Known allergic reaction to cannabis products with previous use
9. Known allergic reaction to sesame oil
10. Known allergic reaction to acetazolamide
11. Pregnant or breast-feeding
12. Current illicit drug abuse (within the last 6 months prior to screening) ; "abuse" has some subsets that are objective and some that require investigator judgement; questions should be discussed with the medical monitor or with the sponsor

    1. An objective subset includes consumption of substances that are "illicit", i.e. not legal per local laws
    2. Investigator judgement is expected for legally marketed products ingested for other than the approved indication(s)
13. Severe depression, defined as a score of ≥30 on the Major Depression Inventory questionnaire
14. Severe anxiety, defined as score of >15 on the General Anxiety Disorder-7 questionnaire
15. Any of the following co-morbid conditions (Note: clarification on co-morbidities and inclusion/exclusion criteria may be discussed with the medical monitor and/or sponsor):

    1. severe psychiatric disorder that might be aggravated or exacerbated by dronabinol's potential to cause anxiety/nervousness, depersonalization, hallucination, etc;
    2. cardiac dysfunction and/or its treatment that might augment dronabinol's potential to cause tachycardia or vasodilation;
    3. marked hepatic dysfunction as defined by elevated ALT or AST >3 times the upper limit of normal, that would reduce dronabinol metabolism; one retest per subject is permitted at the discretion of the investigator; the subject may continue in RePOSA if BOTH repeat transaminase levels are within the reference range;
    4. current or history of encephalopathy or cirrhosis Child-Pugh category B or C (see Appendix 7) since acetazolamide can increase blood ammonia levels precipitating a bout of hepatic encephalopathy;
    5. marked renal dysfunction, including eGFR <60 mL/min/1.73m2, as determined using the National Kidney Foundation calculator
    6. hypokalaemia (low blood potassium), hyponatremia (low blood sodium), hyperchloraemic acidosis, and/or adrenal insufficiency that might be aggravated or exacerbated by acetazolamide's activity as a carbonic anhydrase inhibitor
16. Other ongoing condition(s) that the investigator considers may be clinically significant with regards to the patient's safe participation in this study or may confound this study's findings; any consideration should be discussed with the medical monitor or with the sponsor
17. Participation in any other interventional studies involving investigational or marketed products within 30 days or 5.5 half-lives, whichever is longer, of the IP prior to screening. Patients in Phase II may enter screening (with a different identifier) for Phase III after 30 days from the last administration of the study drug in Phase II.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Estimated)
Dates: Start 2024-05-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in apnea-hypopnea index (AHI) | 4 weeks
  Phase 2 - Assess the change in AHI compared to baseline
Change in apnea-hypopnea index (AHI) | 52 weeks
  Phase 3 - Assess the change in AHI compared to baseline

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Exalt Clinical Research, Chula Vista, California
  - CenExel CNS- Los Alamitos, Long Beach, California
  - Pacific Clinical Research Medical Group, Upland, California
  - Clinical Neuroscience Solutions, Inc. (CNS Healthcare of Jacksonville), Jacksonville, Florida
  - Clinical Neuroscience Solutions, Inc. (CNS Healthcare of Orlando), Orlando, Florida
  - Teradan Clinical Trials, Valrico, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - NeuroTrials Research, Inc., Atlanta, Georgia
  - Tandem Clinical Research, LLC, Marrero, Louisiana
  - Centennial Medical Group, Elkridge, Maryland
  - Meridian Clinical Research, LLC, Rockville, Maryland
  - Henderson Clinical Trials,LLC, Henderson, Nevada
  - Advanced Respiratory and Sleep Medicine, PLLC, Huntersville, North Carolina
  - CTI Clinical Trial and Consulting Services, Cincinnati, Ohio
  - Intrepid Research, Cincinnati, Ohio
  - Velocity Clinical Research - Anderson, Anderson, South Carolina
  - Velocity Clinical Research - Greenville, Greenville, South Carolina
  - Clinical Neuroscience Solutions, Inc. (CNS Healthcare of Memphis), Memphis, Tennessee
  - FutureSearch Trials, Austin, Texas
  - FutureSearch Trials of Dallas, LP, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No